CLINICAL TRIAL: NCT05238480
Title: Effect of Hard Labial Reinforcement of a Custom-made Mouthguard on the Degree of Satisfaction Among Rugby Players. A Randomized Crossover Study
Brief Title: Effect of Hard Labial Reinforcement of a Mouthguard on the Degree of Satisfaction Among Rugby Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Jordi Martinez-Gomis, Associate Professor, Serra Hunter Fellow, Department of Prosthodontics, University of Barcelona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HOUB2021/057
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Satisfaction; Quality of Life
Keywords: Mouthguard; Sports contat
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XC-XP-XP-XC Sequence (Active Comparator): Use of the Xtreme Conventional mouthguard (XC) while playing rugby for first and fourth weeks and the Xtreme Pro mouthguard (XP) for the second and third weeks.
  Interventions: Device: XC mouthguard; Device: XP mouthguard
- XP-XC-XC-XP Sequence (Active Comparator): Use of the Xtreme Pro mouthguard (XP) while playing rugby for first and fourth weeks and the Xtreme Conventional mouthguard (XC) for the second and third weeks.
  Interventions: Device: XC mouthguard; Device: XP mouthguard

INTERVENTIONS:
Device: XC mouthguard — Use of a Xtreme Conventional custom-made mouthguard while playing rugby
Device: XP mouthguard — Use of a Xtreme Pro custom-made mouthguard while playing rugby

SUMMARY:
This study assesses the effect of incorporating a hard labial layer to the front zone of a custom-made mouthguard on the degree of satisfaction of rugby players. Twenty-four rugby players will wear a custom-made Bioplast Xtreme conventional mouthguard (Bioplast Xtreme 4 × 125 + Bioplast 2 x 125; Scheu-Dental Company) and a custom-made Bioplast Xtreme Pro mouthguard (Bioplast Xtreme 4mm × 125 + Duran Layer 0.75mm; Bioplast 2mm x 125), two weeks per mouthguard. They will wear it during training sessions and competitions. The sequence will be randomized for one-half of the participants to start wearing the Bioplast Xtreme conventional and the other half the Bioplast Xtreme Pro mouthguard the first week.

The participants will rate the degree of interference with oral functions or discomfort in reference to speeking, breathing, swallowing, gag reflex, tight or loose fitting, aesthetics and athletic performance, in a 10-point scale, considering 0 no discomfort/interference and 10 maximum discomfort/interference. After each session, players will also rate the perception of the protection, the degree of improvement on athletic performance and the degree of satisfaction in a 10-point scale, considering 0 no protection/satisfaction and 10 maximum protection/satisfaction.

DETAILED DESCRIPTION:
This crossover intervention study aims to assess the effect of incorporating a hard labial layer to the front zone of a custom-made mouthguard on the degree of satisfaction of rugby players. Twenty-four rugby players will participate in this randomized crossover trial. Three hydrocolloid impressions will be made, two of their maxillary arches and one of their mandibular arches, and the casts will be poured immediately with Type IV dental stone. An interocclusal record will be obtained using an extra hard wax covering the tip of two wooden tongue depressors to assure a near centric relation and a minimum interocclusal distance of approximately 2 mm. Two different custom-made mouth guards will be made for each participant, a Bioplast Xtreme conventional mouthguard (Bioplast Xtreme 4 × 125 + Bioplast 2 x 125; Scheu-Dental Company) and a custom-made Bioplast Xtreme Pro mouthguard (Bioplast Xtreme 4mm × 125 + Duran Layer 0.75mm; Bioplast 2mm x 125). Conventional mouthguard will be fabricated using a pressure molding device and a 4-mm ethyl vinyl acetate foil made at 2 mm from the full depth of the labial sulcus, covering the second maxillary molar, and with the palatal margin extending 2 mm from the cervical line. To fabricate the occlusal adjustment a second 2-mm foil of ethyl vinyl acetate will be formed over the initial 4-mm layer. The maxillary and mandibular casts mounted to an articulator using the inter occlusal record will facilitate the accommodation of the occlusal surface to the antagonistic teeth. Bioplast Xtreme Pro will be made by the same procedure, except the incorporation of an extra layer of Duran between 4mm ethyl vinyl acetate foil and 2 mm ethyl vinyl acetate foil. The participants will be instructed to wear the mouth guards during training sessions and competitions. The sequence of use will be randomized to obtain one half of the participants wearing Xtreme Conventional mouthguard the first and the fourth week and the Xtreme Pro mouthguard the second and the third week. The other half will start wearing the first and the fourth week the Xtreme Pro mouthguard and the second and third week the Xtreme conventional mouthguard. The participants will evaluate using a 10-point scale the discomfort (gag reflex, tight or loose fitting), the level of interference with functions (speeking, breathing, swallowing, aesthetics and athletic performance), the protection, and the general satisfaction after each training session or match.

ELIGIBILITY:
Inclusion Criteria:

* Playing in Catalan/Spanish league of rugby for the season 2021-2022

Exclusion Criteria:

* Presence of dental caries
* Players with periodontitis,
* Players with temporomandibular joint pain
* Players with active orthodontic treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Degree of satisfaction using a questionnaire | Weeks 1-4
  Participant satisfaction will be assessed by asking the question "How satisfied are you with your mouthguard?" using a 0-10 point scale, considering 0= totally dissatisfied and 10 = totally satisfied. Players rated the mouthguard just after each training session or after each match.

SECONDARY OUTCOMES:
Degree of interference on speech using a questionnaire | Weeks 1-4
  The degree of interference on speech while using the mouthguard will be assessed by asking the question "How much do you think wearing the mouthguard interferes your ability to speech?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of interference on breathing using a questionnaire | Weeks 1-4
  The degree of interference on breathing while using the mouthguard was assessed by asking the question "How much do you think wearing the mouthguard interferes your ability to breath?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of interference on swallowing using a questionnaire | Weeks 1-4
  The degree of interference on swallowing while using the mouthguard will be assessed by asking the question "How much do you think wearing the mouthguard interferes your ability to swallow?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of discomfort regarding the gag reflex using a questionnaire | Weeks 1-4
  The degree of discomfort regarding the gag reflex while using the mouthguard will be assessed by asking the question "How much do you think wearing the mouthguard causes a gag reflex?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of discomfort because the mouthguard fits too tight using a questionnaire | Weeks 1-4
  The degree of discomfort because the mouthguard fits too tight will be assessed by asking the question "How much do you think the mouthguard fits too tight?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of discomfort related to the dislodgement of the mouthguard using a questionnaire | Weeks 1-4
  The degree of discomfort because the mouthguard dislodges will be assessed by asking the question "How much do you think the mouthguard fits too loose?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of interference on aesthetics using a questionnaire | Weeks 1-4
  The degree of interference on aesthetics while using the mouthguard will be assessed by asking the question "How much do you think wearing the mouthguard interferes on aesthetics?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of interference on athletic performance using a questionnaire | Weeks 1-4
  The degree of interference on athletic performance while using the mouthguard will be assessed by asking the question "How much do you think wearing the mouthguard interferes athletic performance?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of protection using a questionnaire | Weeks 1-4
  The degree of protection perceived by the participant will be assessed by asking the question "How much do you feel protected when you are wearing the mouthguard?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Cost-effectiveness analysis by assessing the degree of satisfaction and the cost of the mouthguard | Weeks 1-4
  The time spent in the laboratory setting and the cost of the materials will be considered for the estimation of the cost-effectiveness of the mouthguard. Effectiveness will be considered as the degree of satisfaction with the mouthguard perceived by the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Martinez-Gomis, DDS PhD, Principal Investigator — University of Barcelona; Jordi Martinez-Gomis, DDS PhD, Study Chair — University of Barcelona
Locations (1):
- Jordi Martinez-Gomis, L'Hospitalet de Llobregat, Catalonia, Spain

REFERENCES:
- [Background] Zamora-Olave C, Willaert E, Montero-Blesa A, Riera-Punet N, Martinez-Gomis J. Risk of orofacial injuries and mouthguard use in water polo players. Dent Traumatol. 2018 Dec;34(6):406-412. doi: 10.1111/edt.12434. Epub 2018 Oct 10. PMID 30156365
- [Background] Gomez-Gimeno A, Zamora-Olave C, Cordobes-Navarro M, Willaert E, Martinez-Gomis J. Satisfaction with shortening the palatal extension of a mouthguard for water polo players: A randomized crossover study. Dent Traumatol. 2019 Apr;35(2):135-141. doi: 10.1111/edt.12455. Epub 2019 Jan 7. PMID 30481393
- [Background] Zamora-Olave C, Willaert E, Parera L, Riera-Punet N, Martinez-Gomis J. Experience with mouthguards and prevalence of orofacial injuries among field hockey players in Catalonia. Dent Traumatol. 2020 Jun;36(3):285-290. doi: 10.1111/edt.12531. Epub 2019 Dec 16. PMID 31765062
- [Background] Flores-Figueiras C, Zamora-Olave C, Willaert E, Martinez-Gomis J. Effect of thickness and occlusal accommodation on the degree of satisfaction with mouthguard use among water polo players: A randomized crossover trial. Dent Traumatol. 2020 Dec;36(6):670-679. doi: 10.1111/edt.12583. Epub 2020 Jul 20. PMID 32590885
- [Background] Iglesias-Porqueras N, Zamora-Olave C, Willaert E, Martinez-Gomis J. Attitudes and opinions towards the prevention of orofacial injuries among water polo coaches in Catalonia: A cross-sectional study. Dent Traumatol. 2021 Aug;37(4):623-630. doi: 10.1111/edt.12675. Epub 2021 Mar 27. PMID 33774914
- [Background] Bochnig MS, Oh MJ, Nagel T, Ziegler F, Jost-Brinkmann PG. Comparison of the shock absorption capacities of different mouthguards. Dent Traumatol. 2017 Jun;33(3):205-213. doi: 10.1111/edt.12324. Epub 2017 Mar 14. PMID 28231638
- [Background] Sarac R, Helbig J, Drager J, Jost-Brinkmann PG. A Comparative Study of Shock Absorption Capacities of Custom Fabricated Mouthguards using a Triangulation Sensor. Materials (Basel). 2019 Oct 28;12(21):3535. doi: 10.3390/ma12213535. PMID 31661939